CLINICAL TRIAL: NCT07296731
Title: Research on Interventions for Anxiety in Cataract Patients Using Preoperative Music Therapy
Brief Title: Anxiety in Cataract Patients Using Preoperative Music Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: k-2025-073-01
Record Dates: First submitted 2025-11-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cataract; Music Therapy
Keywords: Cataract; Music therapy; Preoperative anxiety
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Music therapy (Active Comparator): The patient listened to the selected music through headphones fifteen minutes before the operation.
  Interventions: Behavioral: Music intervention
- Control group (without music therapy) (Placebo Comparator): Patients wore headphones 15 minutes before the operation, but no music was played.
  Interventions: Behavioral: No music intervention

INTERVENTIONS:
Behavioral: Music intervention — Patients listen to the selected music through headphones fifteen minutes before the operation.
  Arms: Experimental:Music therapy
Behavioral: No music intervention — Patients wore headphones 15 minutes before the operation, but no music was played.
  Arms: Control group (without music therapy)

SUMMARY:
The researchers designed this study to investigate whether implementing preoperative music intervention in cataract surgery can reduce perioperative anxiety, alleviate postoperative pain, and enhance patient satisfaction with the surgical procedure.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled single-blind trial. Computer-generated randomization will be used to allocate patients into two groups: a control group (without music therapy) and music therapy group A (listening to music preoperatively). Patient anxiety levels, pain intensity, satisfaction with the surgical procedure, and degree of cooperation during surgery will be assessed through preoperative and postoperative questionnaires and salivary cortisol measurements. Blood pressure and heart rate will be monitored both preoperatively and intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for cataract
* Age ≤ 90 years
* Scheduled for phacoemulsification with IOL implantation under topical anesthesia at the Ophthalmology Department of Guangzhou First People's Hospital
* Voluntarily participates and provides signed informed consent

Exclusion Criteria:

* Requires complex and prolonged surgery, such as:

  1. Shallow anterior chamber with risk of glaucoma
  2. Advanced cataracts with hard nuclei
  3. Small pupils
* Has hearing impairment or communication difficulties
* Shows significant anxiety/depression tendencies or has a history of mental illness with prior/current use of sedatives
* Refuses to participate, or has difficulty understanding/answering questionnaires, or has cognitive impairments
* Uses medications that may affect cortisol and cardiovascular reactivity, including:

  1. Oral contraceptives
  2. Thyroid drugs
  3. Steroids
  4. Psychotropic drugs
* Diagnosed with autoimmune diseases (e.g., Sjögren's syndrome) or oral diseases with inflammation/active lesions

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Salivary Cortisol Levels | Operational day
  Saliva samples were collected at admission and 15 minutes postoperatively using Salivette tubes, centrifuged, and stored at -80°C. Cortisol concentrations were measured via ELISA using the R&D Systems Cortisol Assay Kit (Cat. No. KGE008B)
SATI simplified questionnaire | Operational day
  Anxiety was assessed using the SATI simplified questionnaire (6 items, Likert scale 1-4, 1 = none, 4 = severe)
Visual Analog Scale | Operational day
  Visual Analog Scale (VAS, 0-10, 0 = no anxiety, 10 = extreme anxiety)

SECONDARY OUTCOMES:
Blood pressure | Operational day
  Blood pressure is continuously monitored and recorded in mmHg in the operating room
Intraoperative Pain | Operational day
  Pain intensity was quantified using a VAS (0-10, 0 = no pain, 10 = worst pain)
Heart rate | Operational day
  Heart rate is continuously monitored and recorded in beats per minute in the operating room
Respiratory rate | Operational day
  Respiratory rate is continuously monitored and recorded in breaths per minute in the operating room
The patient's cooperation | Operational day
  The patient's cooperation was assessed by the operating surgeon on a 4-point scale (4=Very Cooperative, 1=Poorly Cooperative).

CONTACTS AND LOCATIONS:
Overall Officials: Yuehong Zhang, Principal Investigator — Guangzhou First People's Hosipital
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangzhou, China